CLINICAL TRIAL: NCT05202678
Title: Prospective, Post-market Evaluation of Safety and Efficacy of a Local Osteo- Enhancement Procedure (LOEP) in the Proximal Femur of Women in Europe with Osteoporosis
Brief Title: RECONFIRM - Study of AGN1 LOEP in Patients with Osteoporosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AgNovos Healthcare, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGN-CIP-301
Record Dates: First submitted 2021-09-23; First posted 2022-01-21 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Osteoporosis
Keywords: Bone mineral density; Femoral strength; Hip fracture; Local osteo-enhancement procedure; LOEP; proximal femur; RECONFIRM
MeSH Terms: conditions — Osteoporosis; Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AGN1 LOEP (Other): Subjects treated with AGN1 LOEP in proximal femur
  Interventions: Device: AGN1 LOEP

INTERVENTIONS:
Device: AGN1 LOEP — Subjects with osteoporosis are treated with AGN1 local osteo-enhancement procedure in the proximal femur

SUMMARY:
The research will be conducted as a prospective, post-market, multi-center study within Europe. The maximum number of subjects to be treated is 150 across up to 20 sites. This will be a non-randomized and open-label study. The study will collect procedural, short- and long-term data on the safety and clinical performance of AGN1 LOEP in the post-market setting in European countries where AGN1 LOEP is commercially available. AGN1 is intended to form new bone in voids in the proximal femur of women with osteoporosis.

DETAILED DESCRIPTION:
To qualify for this study, a subject must have at least one intact hip with bone loss attributable to osteoporosis as indicated by a femoral neck DXA T-score of -2.5 or less.

Follow-up visits will be conducted at 10 days, 42 days, 12 months, and 24 months after the procedure. Study evaluations at each follow-up visit include general health (physical exam and medical history update), VAS pain (not at 10 days), FES-I (not at 10 days), EQ5D-5L and Parker Mobility. A Timed Up and Go Test is performed at the 10-day, 42-day and 12-month follow-up. Patient satisfaction with outcome of surgery will be asked at the 42-day and the 12-month follow-up. DXA scans and X-rays will be performed at 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a postmenopausal female (at least 1-year post menses).
2. Subject has bone loss in the hip attributable to osteoporosis as defined by a femoral neck DXA T-score of -2.5 or less.
3. Subject has at least one hip without previous surgery or fracture.
4. Subject is medically stable from any previous treatment or medical procedure in the opinion of the investigator and with an ASA score of I or II.
5. Subject has willingness, ability, and commitment to participate in baseline and follow-up evaluations for the full length of the study.
6. Subject is capable of giving written informed consent to participate in the study.

Exclusion Criteria:

1. Subject is less than 3 months removed from having a hip fracture repair or prosthesis or elective Total Hip Arthroplasty (THA).
2. Subject has progressive increase in hip pain over the previous six (6) months that in the opinion of the Investigator suggests moderate to severe intra-articular arthritis, labral tear, extraarticular soft tissue pathology, referred pain, tumor, stress fracture or infection.
3. Subject is dependent on the use of a wheelchair or is bedridden.
4. Subject has albumin corrected serum calcium levels outside the normal lab range or has a pre-existing calcium metabolism disorder (e.g., hypercalcemia).
5. Subject has severe renal insufficiency defined as an estimated glomerular filtration rate (eGFR) < 30 mL/min or is being treated with dialysis.
6. Subject has hemoglobin A1c level ≥ 7.5%.
7. Subject has Body Mass Index (BMI) > 35.
8. Subject exhibits excessive smokeless tobacco use or excessive smoking as determined by the principal investigator*.
9. Subject is at ASA Class III, IV, V or VI.
10. Subject exhibits excessive alcohol consumption as determined by the principal investigator*.
11. Subject has radiological evidence of gross bony or joint pathology of the hip, including signs predictive of atypical femoral fractures (e.g., Cortical beaking) or has been diagnosed and/or treated for atypical femoral fractures.
12. Subject treated with corticosteroids or systemic glucocorticoids for ten (10) days in the previous six (6) months.
13. Subject has history of oral or parenteral use of immunesuppressive drugs in the previous twelve months.
14. Subject has history of metabolic bone disease other than osteoporosis (ex. Paget's disease).
15. Subject has a history of auto-immune arthritic diseases including rheumatoid, psoriatic, or those associated with systemic lupus erythematosus, spondyloarthropathy, Reiter's Syndrome or Crohn's Disease.
16. Subject has a history of radiation therapy to the hip or pelvic region.
17. Subject has a history of any invasive malignancy (except basal cell carcinoma), unless treated and with no clinical signs or symptoms of the malignancy for five (5) years.
18. Subject has known allergies to implanted device.
19. In the judgement of the Investigator, the subject is not a good study candidate (e.g., inability to maintain follow-up schedule, comorbidity or poor general physical/mental health, or drug or alcohol abuse issues).
20. Subject is currently enrolled in another clinical study. *AgNovos's recommendation is >1 pack per day smoking and >3 alcoholic drinks per day

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Postmenopausal female with a femoral neck T-score of 2.5 or less
Enrollment: 150 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Femoral Neck Bone Mineral Density | 12 months
  6% increase in mean femoral neck BMD from preprocedure baseline to 12 months post-procedure of treated hips
Primary Safety Evaluation | 12 months
  The incidence of all adverse events and serious adverse events occurring post-AGN1 LOEP through the 12 months follow-up period determined to be at least possibly related to the procedure and/or device.

SECONDARY OUTCOMES:
Total Hip Bone Mineral Density | 12 months
  6% increase in mean total hip BMD from preprocedure baseline to 12 months post-procedure of treated hips.
Femoral Neck Bone Mineral Density | 24 months
  6% increase in mean femoral neck BMD from preprocedure baseline to 24 months post-procedure of treated hips.
Total Hip Bone Mineral Density | 24 months
  6% increase in mean total hip BMD from preprocedure baseline to 24 months post-procedure of treated hips.

OTHER OUTCOMES:
Bone Formation | 12 and 24 months
  Radiologic appearance of bone formation as assessed by X-ray at 12 and 24 months post-procedure of treated hips.
Patient Satisfaction | 42 days and 12 months
  Patient satisfaction with outcome of surgery in the treated hip(s) and overall at 42 days and 12 months assessed with Visual Analogue Scale.
Pain hip | baseline, 42 days, 12 months, and 24 months.
  Pain (left hip, right hip) at baseline, 42 days, 12 months, and 24 months assessed with Visual Analogue Scale.
Pain body overall | baseline, 42 days, 12 months, and 24 months.
  Pain body overall at baseline, 42 days, 12 months, and 24 months assessed with Visual Analogue Scale.
FES-I | baseline, 42 days, 12 months, and 24 months
  FES-I at baseline, 42 days, 12 months, and 24 months
Quality of Life with EQ5D-5L | baseline, 10 days, 42 days, 12 months, and 24 months
  EQ5D-5L at baseline, 10 days, 42 days, 12 months, and 24 months
Parker Mobility Score | baseline, 10 days, 42 days, 12 months, and 24 months.
  Parker Mobility Score at baseline, 10 days, 42 days, 12 months, and 24 months.
Verifying the enhancement site | Procedure (day 0)
  The ability to access the enhancement site by drilling through the lateral femoral cortex of the proximal femur and to determine the boundaries of the enhancement site using the probe debrider.
Technical Success | Procedure (day 0)
  The ability to deliver the necessary amount of AGN1 material to adequately fill the osseous defect as assessed by the treating surgeon.
SAE | 24 months
  Incidence of all serious adverse events post-AGN1 LOEP through the 24 months follow-up period.
Hip Fracture | 24 months
  Incidence of new hip fractures on the treated side.
Timed up and go test | baseline, 10 days, 42 days and 12 months.
  Timed up and go test at baseline, 10 days, 42 days and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jo De Schepper, MD, Principal Investigator — AZ Nikolaas
Locations (1):
- AZ Nikolaas, Sint-Niklaas, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: No